CLINICAL TRIAL: NCT00264212
Title: A Multicentre Prospective Randomized Open-Label 12-Week Study With Blinded Evaluation Comparing the Efficacy and Safety of Irbesartan and Irbesartan-Hydrochlorothiazide Fixed Combination With Amlodipine and Amlodipine Plus Hydrochlorothiazide in Elderly Patients With Isolated Systolic Hypertension
Brief Title: AMISH : Aprovel for Management of Isolated Systolic Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R_8791
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

INTERVENTIONS:
Drug: irbesartan and irbesartan-hydrochlorothiazide

SUMMARY:
To compare the antihypertensive efficacy and tolerability of irbesartan and irbesartan-hydrochlorothiazide fixed combination therapy with amlodipine and amlodipine plus hydrochlorothiazide in the treatment of isolated systolic hypertension.

ELIGIBILITY:
Main criteria are listed hereafter:

Inclusion Criteria:

* at Screening

  * Outpatients
  * With newly diagnosed and untreated OR previously diagnosed, treated and uncontrolled Isolated Systolic Hypertension defined as:

    * seated Systolic Blood Pressure (SBP) ≥ 160mmHg and < 220 mmHg [160-220[
    * AND seated Diastolic Blood Pressure (DBP)< 90 mmHg
* at Randomization

  * Having completed the 2 to 4-week wash-out/placebo run-in phase
  * Still eligible for Blood Pressure
  * seated SBP ≥ 160mmHg and < 220 mmHg [160-220[
  * AND seated DBP < 90 mmHg.

Exclusion Criteria (at Screening):

* Participation in a clinical trial within the previous 3 months
* Patients with a history of irbesartan, amlodipine, or hydrochlorothiazide sensitivity defined as irbesartan, amlodipine, or hydrochlorothiazide discontinuation due to medically significant adverse effects
* Patients currently or previously treated with Angiotensin II Receptor Blocker (irbesartan, losartan, candesartan, valsartan, telmisartan, etc.) or dihydropiridine Calcium Channel Blocker (amlodipine, nicardipine, felodipine, nifedipine, etc.) AND not responding despite maximum tolerated dose
* Known or suspected secondary hypertension (e.g., coarctation of aorta, renovascular stenosis, etc.)
* Known single functional kidney
* History of recent myocardial infarction, coronary artery bypass graft surgery or percutaneous transluminal coronary angioplasty, or cerebrovascular accident (Transient Ischaemic Attack, stroke) within the last 6 months of study entry
* Patients with known gastrointestinal, renal, hepatic, endocrine, cardiovascular, pulmonary, immunological or hematological disease which in the opinion of the investigator is active or uncontrolled
* Patients with significant renal (clearance of creatinine < 30 mL/mn), hepatic or cardiac insufficiency, or known valvular heart disease
* Serum potassium < 3.5 mmol/L (mEq/L) or > 5.5 mmol/L (mEq/L)
* Presence of clinically significant ventricular or supraventricular arrhythmias, or second or third degree atrioventricular block, or QTc prolongation (Bazett > 450 msec.) on the ECG
* Pregnancy or lactation. Women of child bearing potential (not post-menopausal) should be using a reliable contraceptive method

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436
Dates: Start 2004-08

PRIMARY OUTCOMES:
Change from baseline in office seated SBP at week 12

SECONDARY OUTCOMES:
At 4, 8 and 12 weeks: Number of responders and normalized, Change from baseline in pulse pressure (SBP-DBP), Change from baseline in standing SBP, Safety : Change in standing SBP/DBP, incidence of orthostatic hypotension, adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pascale BLONDIN, MD, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis, Santiago, Chile
- Sanofi-Aventis, Shanghai, China
- Sanofi-Aventis, Jakarta, Indonesia
- Sanofi-Aventis, México, Mexico
- Sanofi-Aventis, Manila, Philippines
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-Aventis, Taipei, Taiwan
- Sanofi-Aventis, Bangkok, Thailand